CLINICAL TRIAL: NCT05617807
Title: Outcomes of the Nanoscopic Partial Meniscectomy Versus Standard Arthroscopic Partial Meniscectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall University (Other)
Collaborators: Arthrex, Inc. (Industry); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Shane Taylor, Principal Investigator, Marshall University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1926751-2
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Meniscus Tear
Keywords: Arthroscopy; Meniscus; Meniscectomy; Nanoscopic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Nanoscopic Partial Meniscectomy (Experimental): This is the experimental group. patients will have a partial meniscectomy performed using the arthrex nanoscope
  Interventions: Procedure: Nanoscopic partial meniscectomy
- Standard Partial Meniscectomy (Active Comparator): Patients will have a partial meniscectomy performed using standard arthroscopic equipment which is the current gold standard
  Interventions: Procedure: Standard Partial Meniscectomy

INTERVENTIONS:
Procedure: Nanoscopic partial meniscectomy — Patients will have a partial meniscectomy performed using the arthrex nanoscope and it will be compared to partial meniscectomy performed using standard arthroscopic equipment
  Arms: Nanoscopic Partial Meniscectomy
Procedure: Standard Partial Meniscectomy — Patients will have partial meniscectomy performed using standard arthroscopic equipment
  Arms: Standard Partial Meniscectomy

SUMMARY:
Standard arthroscopy has been the gold standard for treatment of meniscus tears since the 1980's. The purpose of this study is to analyze the clinical outcomes of using the smaller diameter Nanoscope for partial menisectomy. The authors hypothesize that the Nanoscopic partial menisectomy patients will have less pain and return function faster than standard arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* MRI positive for meniscus tear
* More than 3mm of joint space on PA flexion weightbearing x rays
* Primary arthroscopy

Exclusion Criteria:

* Workers compensation
* Older than 60 years of age
* Revision surgeries

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Functional Outcomes following partial meniscectomy: Knee Injury and Osteoarthritis Score | 6 weeks
  We will be looking at functional outcomes following partial meniscectomy with the nanoscope compared to standard arthroscopy by looking at Knee Injury and Osteoarthritis Score (O -100 with higher being patients doing better functionally)
Functional Outcomes Following Partial Meniscectomy: International Knee Documentation Committee Score | 6 weeks
  We will be looking at functional outcomes following partial meniscectomy with the nanoscope compared to standard arthroscopy by looking at the International Knee Documentation Committee Score (0-100 with higher being patients doing better functionally)

SECONDARY OUTCOMES:
Pain: Visual Analog Pain Score | 6 weeks
  Pain following partial meniscectomy with the nanoscope compared to standard arthroscopy using Visual Analog Pain Score (0-10 with 0 being no pain and 10 being the worst pain)
Narcotic Medication Use | 24 hours
  we will be looking at the amount of narcotic pain medication used following nanoscopic partial meniscectomy compared to standard arthroscopy
Return to work | 6 weeks
  time to return to work following partial meniscectomy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Marshall Orthopaedics - Teays Valley, Scott Depot, West Virginia

IPD SHARING:
Plan to Share IPD: No